CLINICAL TRIAL: NCT05325008
Title: An Adaptive Randomised Controlled Trial to Treat Polyomavirus Infections (BKPyV) in Kidney and Kidney Pancreas Transplant Recipients
Brief Title: A Trial to Treat Polyomavirus Infections (BKPyV) in Kidney and Simultaneous Kidney Pancreas Transplant Recipients
Acronym: BEAT-BK
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Queensland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AKTN 20.07
Record Dates: First submitted 2022-01-10; First posted 2022-04-13 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-10

CONDITIONS: BK Viremia; Kidney Transplant Infection; Kidney Transplant Failure and Rejection
Keywords: Kidney transplantation; Intravenous immunoglobulin; Virus; Nephropathy; Clinical trial; Nephrology
MeSH Terms: conditions — Rejection, Psychology; Virus Diseases; Kidney Diseases | interventions — Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Immunosuppression reduction/modification + Intravenous Immunoglobulin (Experimental): Receives Immunosuppression reduction/modification + Intravenous Immunoglobulin
  Interventions: Drug: Immunosuppression reduction/modification + intravenous immunoglobulin
- Immunosuppression reduction/modification (Other): Receives Immunosuppression reduction/modification as part of standard of care.
  Interventions: Other: Immunosuppression reduction/modification

INTERVENTIONS:
Drug: Immunosuppression reduction/modification + intravenous immunoglobulin — Participants will receive intravenous immunoglobulin along with immunosuppression reduction/modification.
  Other Names: Human immunoglobulin
  Arms: Immunosuppression reduction/modification + Intravenous Immunoglobulin
Other: Immunosuppression reduction/modification — Participants will receive immunosuppression reduction/modification.
  Arms: Immunosuppression reduction/modification

SUMMARY:
BEAT-BK will see the effect of immunosuppression reduction/modification with and without IVIG on BKPyV infection, allograft function, allograft loss, acute transplant rejection, immunosuppression load and death in kidney and simultaneous kidney pancreas transplant recipients with polyomavirus infections (BKPyV).

DETAILED DESCRIPTION:
BKPyV infection is a rare but also devastating disease in kidney and SPK transplant recipients. Immunosuppression used in transplantation minimises the risk of acute rejection and eventual graft loss, but suppression of the immune system increases the risk of opportunistic infections and reactivation of latent viruses causing disease, such as BKPyV infection. Therefore, balancing the complications of excessive versus inadequate immunosuppression is a key priority for patients and health professionals. The BEAT-BK trial is designed through a structured, consensus process, and informed by the pilot observational data generated by the investigators. The conventional immunosuppression reduction approach may include judicious reduction in the doses of calcineurin inhibitors and anti-proliferative agents, or conversion to less potent immunosuppression therapy such as a switch from tacrolimus to cyclosporine, or mycophenolate to azathioprine. While adjuvant therapy is not commonly used, 63% of participants would consider IVIG as a 'rescue', when conventional therapy has failed, or the graft function is deteriorating rapidly. IVIG is a nondepleting agent containing natural antibodies with potential antiviral and immunomodulatory properties. It is used against some chronic infections (Epstein-Barr virus) and the treatment of antibody-mediated rejection in kidney transplantation. In BKPyV infection, the certainty of the evidence for IVIG is very low due to imprecision, and high risk of bias (small, case series, retrospective cohorts), but it holds promise based on findings from our observational data (n = 50). Recipients with BKPyV-DNAemia who received IVIG as adjuvant therapy were more likely to achieve complete viral clearance at 12 months (77.3% vs. 33.3%, p < 0.01) and less likely to relapse (11% vs. 27.3%, p=0.01) compared to recipients who received conventional therapy alone.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 2 years or above
2. Have received a kidney or simultaneous pancreas-kidney transplant
3. Have BKPyV-Viremia (detected by RT-PCR) with a viral count ≥ 5,000 copies per mL, or histological confirmation of BKPyVAN, within 3 weeks prior to randomisation.
4. Be able to provide informed consent or consent given by a parent or guardian (if age <18 years) or other authorised person

Exclusion Criteria:

1. Contraindications to receiving IVIG as a treatment
2. Current active acute rejection (≤ 3 months prior)
3. Treating clinicians would regard as unsafe to be enrolled
4. Limited life expectancy (< 12 months)
5. Receiving Belatacept as part of their immunosuppression protocol
6. Currently undergoing or who have previously received, viral-specific T-cell therapy for BK viremia
7. Prior infection and treatment for BKPyV-Viremia
8. Received IVIG treatment in the past with last IVIG treatment < 4 weeks prior to randomisation

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 280 (Estimated)
Dates: Start 2023-08-18 (Actual); Primary Completion 2027-08-01 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Composite ordinal outcome based on all cause death, allograft loss, eGFR decline, acute allograft rejection or BKV load > 1000 copies/mL, and immunosuppression load. | 11 - 13 weeks
  All participants will be allocated a rank at 12 weeks between rank 5 (worst) and rank 1 (best). The primary comparison of interest is between participants randomised to intravenous immunoglobulin (IVIG) and participants randomised to the control arm.
  Outcome measures include: Rank 5 - all cause death, allograft loss, eGFR decline ≥10mls/min 1.73². Rank 4 - acute allograft rejection or BK viral load to >1000 copies/mL. Ranks 3, 2, and 1 - the degree of immunosuppression reduction relative to baseline immunosuppression.

SECONDARY OUTCOMES:
BKPyV final viral load | 12 weeks
  Compare the number of participants in the intervention and control groups with a BK Polyomavirus viral load to <1000 copies/mL
eGFR decline | 12, 24 & 48 weeks
  Compare the number of participants in the intervention and control groups with an estimated glomerular filtration rate (eGFR) decline ≥ 10 ml/min/1.73 m2
All cause death | 12, 24 & 48 weeks
  Compare the mortality rate in the intervention and control groups.
Graft loss | 12, 24 & 48 weeks
  Compare the number of graft survival and death-censored graft survival participants in the intervention and control groups.
Acute rejection of kidney and/or pancreas allografts | 12 & 48 weeks
  Compare the number of acute rejections (cellular and antibody mediated) episodes between the intervention and control groups.
Donor Specific Anti-HLA Antibody | 12 & 48 weeks
  Compare the number of participants that develop de novo donor-specific antibodies between the intervention and control groups
Infusion reactions and/ or venous thromboembolism events | 12 weeks
  Compare the incidence rate (number) of infusion reactions and venous thromboembolism between the intervention and control groups
Hospitalisations due to infection events | Baseline,1,2,3,4,5,6,7,8,10,12,24,48 weeks
  Compare the number of hospitalisation due to infection between the intervention and control groups.
Number of infectious events requiring antimicrobial (antibacterial, antiviral, antifungal, antiprotozoal) therapy. | Baseline,1,2,3,4,5,6,7,8,10,12,24,48 weeks
  Compare the number of infectious events requiring antimicrobial therapy between the intervention and control groups
EuroQol-5 Dimension-5 Level for adults/ Health Utilities Index-3 for children | Baseline, 12, 24 & 48 weeks
  Compare the outcomes of health-related quality of life between the intervention and control groups.
BK polyomavirus associated nephropathy events | 12 & 48 weeks
  Compare the number of participants that develop BK polyomavirus associated nephropathy between the intervention and control groups
Any cancer diagnosis or cancer related death | 24 & 48 weeks
  Compare the incidence rate (number) of cancer outcomes between the intervention and control groups.
Composite ranked outcome | 24 & 48 weeks
  Compare the long-term composite ranked outcome between the intervention and control groups
Adverse events of special interest and serious adverse events | Baseline,1,2,3,4,5,6,7,8,10,12,24,48 weeks
  Compare the incidence rate (number) of safety related events between intervention and control group.

CONTACTS AND LOCATIONS:
Overall Officials: Germaine Wong, Professor, Study Chair — University of Sydney
Locations (12):
- Australia (12):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - John Hunter Hospital, New Lambton Heights, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal Prince Alfred Hospital, Sydney, New South Wales
  - The Childrens Hospital Westmead, Sydney, New South Wales
  - Western Sydney Local Health District (Westmead Hospital), Westmead, New South Wales
  - Queensland Children's Hospital, Brisbane, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Flinders Medical Centre, Adelaide, South Australia
  - Monash Health, Melbourne, Victoria
  - Perth Children's Hospital, Perth, Western Australia
  - Sir Charles Gairdner Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Helle F, Aubry A, Morel V, Descamps V, Demey B, Brochot E. Neutralizing Antibodies Targeting BK Polyomavirus: Clinical Importance and Therapeutic Potential for Kidney Transplant Recipients. J Am Soc Nephrol. 2024 Oct 1;35(10):1425-1433. doi: 10.1681/ASN.0000000000000457. Epub 2024 Jul 9. PMID 39352862